CLINICAL TRIAL: NCT00001019
Title: A Phase I Clinical Trial to Evaluate:Part A. The Safety and Immunogenicity of Two Dose Levels of SF-2 gp120 (CHO) With or Without MTP-PE Adjuvant in the MF59 Emulsion Part B. The Safety and Immunogenicity of Five Monthly Doses of 50 mcg gp120 Protein in MF59 Emulsion (Without MTP-PE) Versus the Emulsion Control
Brief Title: Safety of and Immune Response to an HIV Vaccine (SF-2 gp120) With or Without MTP-PE/MF59 Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 007A/B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Adjuvants, Immunologic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1 SF-2
Biological: MTP-PE/MF59

SUMMARY:
Part A: To compare the safety and immunogenicity of two dose levels of gp120 (CHO) in MF59 emulsion alone or with MTP-PE/MF59 adjuvant, administered at 0, 1, and 6 months.

Part B: To evaluate the safety and immunogenicity of gp120 in MF59 when administered in five monthly injections.

One experimental AIDS vaccine is the gp120 vaccine. The HIV envelope glycoprotein 120 is manufactured through recombinant DNA technology and used as an immunogen. Antibodies directed against gp120 can neutralize HIV-1, and gp120 can also stimulate certain types of cell-mediated immune responses. Because many immunogens, including candidate HIV vaccines, may evoke relatively weak immune responses, the use of adjuvants, or substances that augment immune responses to vaccines, is of interest. MTP-PE/MF59, composed of the immunomodulator MTP-PE combined with MF59 emulsion, appears to be a promising adjuvant and has been selected for studies with the gp120 vaccine.

DETAILED DESCRIPTION:
One experimental AIDS vaccine is the gp120 vaccine. The HIV envelope glycoprotein 120 is manufactured through recombinant DNA technology and used as an immunogen. Antibodies directed against gp120 can neutralize HIV-1, and gp120 can also stimulate certain types of cell-mediated immune responses. Because many immunogens, including candidate HIV vaccines, may evoke relatively weak immune responses, the use of adjuvants, or substances that augment immune responses to vaccines, is of interest. MTP-PE/MF59, composed of the immunomodulator MTP-PE combined with MF59 emulsion, appears to be a promising adjuvant and has been selected for studies with the gp120 vaccine.

In Part A, 32 volunteers (eight on each of four treatment arms) are randomized to receive one of two doses (15 or 50 mcg) of gp120 vaccine with either MTP-PE/MF59 adjuvant emulsion or MF59 emulsion alone. The volunteers receive three IM injections at 0, 1, and 6 months. In Part B, 16 female volunteers (eight on each of two treatment arms) are randomized to receive either MF59 emulsion alone (placebo) or MF59 emulsion plus gp120 vaccine (50 mcg). Volunteers receive five IM injections at monthly intervals.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Normal history and physical exam.
* No identifiable high-risk behavior for HIV infection.
* Negative ELISA for HIV.
* Normal cell-mediated immune responses using Merieux skin test.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant evidence of depression.
* Positive syphilis serology (e.g., RPR) that is documented not to be a false positive or from a remote (> 6 months) treated infection.
* Circulating Hepatitis B antigenemia.
* More than two sexual partners, or sexual contact with a high-risk partner, within the past 6 months.

Patients with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* Significant evidence of depression or under treatment for psychiatric problems within the past year.
* History of anaphylaxis or other adverse vaccine reactions.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) within the past 6 months.

Prior Medication:

Excluded:

* Immunoglobulin or vaccines within the past 2 months.
* Experimental agents within the past 30 days.

Prior Treatment:

Excluded:

* Blood transfusions or cryoprecipitates within the past 3 months.

Risk Behavior: Excluded:

* History of IV drug use within the past year.
* More than two sexual partners, or sexual contact with a high-risk partner, within the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Overall Officials: Graham B, Study Chair
Locations (4):
- United States (4):
  - St Louis Univ School of Medicine, St Louis, Missouri
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Univ Hosp, Nashville, Tennessee
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington

REFERENCES:
- [Background] Graham BS, Keefer MC, McElrath MJ, Gorse GJ, Schwartz DH, Weinhold K, Matthews TJ, Esterlitz JR, Sinangil F, Fast PE. Safety and immunogenicity of a candidate HIV-1 vaccine in healthy adults: recombinant glycoprotein (rgp) 120. A randomized, double-blind trial. NIAID AIDS Vaccine Evaluation Group. Ann Intern Med. 1996 Aug 15;125(4):270-9. doi: 10.7326/0003-4819-125-4-199608150-00003. PMID 8678389
- [Background] Kahn JO, Sinangil F, Baenziger J, Murcar N, Wynne D, Coleman RL, Steimer KS, Dekker CL, Chernoff D. Clinical and immunologic responses to human immunodeficiency virus (HIV) type 1SF2 gp120 subunit vaccine combined with MF59 adjuvant with or without muramyl tripeptide dipalmitoyl phosphatidylethanolamine in non-HIV-infected human volunteers. J Infect Dis. 1994 Nov;170(5):1288-91. doi: 10.1093/infdis/170.5.1288. PMID 7963729